CLINICAL TRIAL: NCT05128058
Title: AN OPEN LABEL, PHASE 1, TWO-ARM STUDY TO ASSESS TARGET OCCUPANCY AND FUNCTIONAL INHIBITION OF JAK3 AND TEC KINASES BY SINGLE DOSES OF RITLECITINIB IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Target Occupancy Study With Ritlecitinib.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B7981045
Record Dates: First submitted 2021-10-15; First posted 2021-11-19 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Subjects will be dosed with 50 mg Ritlecitinib on Day 1 and followed up till Day 3
  Interventions: Drug: Ritlecitinib 50 mg
- Cohort 2 (Experimental): Subjects will be dosed with 200 mg Ritlecitinib on Day 1 and followed up till Day 3
  Interventions: Drug: Ritlecitinib 200 mg

INTERVENTIONS:
Drug: Ritlecitinib 50 mg — 50 mg single dose
  Other Names: PF-06651600
  Arms: Cohort 1
Drug: Ritlecitinib 200 mg — 200 mg single dose
  Other Names: PF-06651600
  Arms: Cohort 2

SUMMARY:
This is a phase 1, open label, two-arm study to assess target occupancy and functional inhibition of JAK3 and TEC kinases by Ritlecitinib in healthy adult participants

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination including BP and pulse rate measurement, 12-lead ECG, or clinical and laboratory tests.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Infection with HIV, hepatitis B or hepatitis C viruses
* Have evidence of untreated or inadequately treated active or latent Mycobacterium TB infection
* Known active or history of recurrent bacterial, viral, fungal, mycobacterial or other infections.
* Have received only one of the 2 required doses of COVID-19 vaccine.
* Participants have a known present or a history of malignancy other than a successfully treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Saadeddin A, Purohit V, Huh Y, Wong M, Maulny A, Dowty ME, Sagawa K. Virtual Bioequivalence Assessment of Ritlecitinib Capsules with Incorporation of Observed Clinical Variability Using a Physiologically Based Pharmacokinetic Model. AAPS J. 2024 Jan 24;26(1):17. doi: 10.1208/s12248-024-00888-9. PMID 38267790
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981045

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 participants were assigned to study treatment; 8 in the ritlecitinib 50 mg group and 8 in the ritlecitinib 200 mg group. All the participants were treated in this study.
Groups:
- RITLECITINIB 50 MG CAPSULE: Healthy participants enrolled to receive 50 mg single dose of ritlecitinib capsule on Day 1.
- RITLECITINIB 200 MG CAPSULE: Healthy participants enrolled to receive 200 mg single dose of 4 ritlecitinib 50 mg capsules on Day 1.
Period: Overall Study
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (10.95) | 37.9 (12.97) | 40.9 (12.0)
Age, Customized [Number; unit: Participants]
  <18 | 0 | 0 | 0
  18-44 | 3 | 4 | 7
  45-64 | 5 | 4 | 9
  >=65 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 4 | 4 | 8
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Target Occupancy for JAK3
Description: Target occupancy for janus kinase 3 (JAK3) in peripheral blood mononuclear cells (PBMCs) by ritlecitinib was investigated in human blood by chemical probe-based enrichment and liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS) analysis. % TO is calculated as [(baseline value - value at specified time point)*100/baseline value], where baseline value in this formula is defined as the mean of the two pre-dose measurements at Hour -1 and Hour 0 on Day 1. Since (baseline value - value at specified time point)=0 at baseline, % TO at baseline is 0.
Time Frame: -1 (pre-dose), 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: The analysis population included all participants who enrolled and treated with non-misssing value at the specified time point.
Measure: Median (Full Range); unit: percentage of occupancy
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
percentage of occupancy
  Baseline | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]
  1H | 72.41 [49.2 to 98.0] | 28.74 [-5.8 to 51.1]
  2H | 12.28 [-30.1 to 39.5] | 64.14 [54.1 to 75.0]
  4H | -1.39 [-19.6 to 5.2] | 62.06 [45.3 to 73.9]
  8H | -23.34 [-49.1 to 17.7] | 58.76 [38.9 to 65.2]
  24H | -24.72 [-58.2 to -10.2] | 37.08 [30.2 to 53.1]
  48H | -25.34 [-51.8 to 3.7] | 33.44 [9.4 to 52.9]

2. Primary Outcome: Percent Target Occupancy for BTK
Description: Target occupancy for Bruton's tyrosine kinase (BTK) in PBMCs by ritlecitinib was investigated in human blood by chemical probe-based enrichment and LC-MS/MS analysis. % TO is calculated as [(baseline value - value at specified time point)*100/baseline value], where baseline value in this formula is defined as the mean of the two pre-dose measurements at Hour -1 and Hour 0 on Day 1. Since (baseline value - value at specified time point)=0 at baseline, % TO at baseline is 0.
Time Frame: -1 (pre-dose), 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of occupancy
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
percentage of occupancy
  Baseline | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]
  1H | 98.45 [95.4 to 99.8] | 99.57 [98.2 to 99.8]
  2H | 96.83 [92.1 to 99.2] | 99.37 [98.6 to 99.8]
  4H | 96.43 [90.4 to 99.1] | 99.35 [99.2 to 99.8]
  8H | 93.52 [85.3 to 97.8] | 99.21 [97.1 to 99.5]
  24H | 83.21 [76.5 to 86.3] | 92.13 [87.0 to 95.5]
  48H | 69.86 [63.3 to 76.4] | 82.66 [75.8 to 88.1]

3. Primary Outcome: Percent Target Occupancy for ITK
Description: Target occupancy forIL 2 inducible T-cell kinase (ITK) in PBMCs by ritlecitinib was investigated in human blood by chemical probe-based enrichment and LC-MS/MS analysis. % TO is calculated as [(baseline value - value at specified time point)*100/baseline value], where baseline value in this formula is defined as the mean of the two pre-dose measurements at Hour -1 and Hour 0 on Day 1. Since (baseline value - value at specified time point)=0 at baseline, % TO at baseline is 0.
Time Frame: -1 (pre-dose), 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of occupancy
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
percentage of occupancy
  Baseline | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]
  1H | 94.40 [86.2 to 100.0] | 97.03 [73.8 to 98.0]
  2H | 67.77 [42.2 to 88.4] | 97.06 [94.5 to 98.1]
  4H | 57.54 [23.0 to 73.9] | 92.27 [86.0 to 97.4]
  8H | 28.76 [-5.5 to 58.0] | 76.59 [60.0 to 88.9]
  24H | -16.77 [-42.1 to 30.5] | 32.33 [12.4 to 43.8]
  48H | -9.87 [-61.0 to 21.6] | 20.62 [-16.0 to 44.7]

4. Primary Outcome: Percent Target Occupancy for TXK
Description: Target occupancy for tyrosine kinase expressed in T cells (TXK) in PBMCs by ritlecitinib was investigated in human blood by chemical probe-based enrichment and LC-MS/MS analysis. % TO is calculated as [(baseline value - value at specified time point)*100/baseline value], where baseline value in this formula is defined as the mean of the two pre-dose measurements at Hour -1 and Hour 0 on Day 1. Since (baseline value - value at specified time point)=0 at baseline, % TO at baseline is 0.
Time Frame: -1 (pre-dose), 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of occupancy
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
percentage of occupancy
  Baseline | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]
  1H | 100.00 [88.6 to 100.0] | 100.00 [37.7 to 100.0]
  2H | 44.97 [27.1 to 66.7] | 100.00 [100.0 to 100.0]
  4H | 34.01 [-15.8 to 52.1] | 100.00 [87.9 to 100.0]
  8H | 23.17 [-41.0 to 60.7] | 82.46 [63.1 to 100.0]
  24H | -4.09 [-43.4 to 31.4] | 49.70 [33.2 to 59.7]
  48H | -38.98 [-83.7 to 17.7] | 20.34 [1.9 to 58.8]

5. Primary Outcome: Percent Target Occupancy for TEC
Description: Target occupancy for tyrosine kinase expressed carcinoma (TEC) in PBMCs by ritlecitinib was investigated in human blood by chemical probe-based enrichment and LC-MS/MS analysis. % TO is calculated as [(baseline value - value at specified time point)*100/baseline value], where baseline value in this formula is defined as the mean of the two pre-dose measurements at Hour -1 and Hour 0 on Day 1. Since (baseline value - value at specified time point)=0 at baseline, % TO at baseline is 0.
Time Frame: -1 (pre-dose), 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of occupancy
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
percentage of occupancy
  Baseline | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]
  1H | 96.50 [87.4 to 100.0] | 100.0 [96.0 to 100.0]
  2H | 94.60 [88.3 to 98.0] | 99.42 [98.3 to 100.0]
  4H | 94.23 [90.9 to 98.3] | 98.78 [98.1 to 100.0]
  8H | 93.12 [85.5 to 98.6] | 99.57 [97.4 to 100.0]
  24H | 90.64 [83.7 to 95.8] | 96.85 [94.1 to 97.8]
  48H | 82.48 [75.7 to 87.3] | 92.32 [87.9 to 94.8]

6. Primary Outcome: Percent Target Occupancy for BMX
Description: Target occupancy for bone marrow tyrosine kinase gene in chromosome X (BMX) in PBMCs by ritlecitinib was investigated in human blood by chemical probe-based enrichment and LC-MS/MS analysis. % TO is calculated as [(baseline value - value at specified time point) *100/baseline value], where baseline value in this formula is defined as the mean of the two pre-dose measurements at Hour -1 and Hour 0 on Day 1. Since (baseline value - value at specified time point)=0 at baseline, % TO at baseline is 0.
Time Frame: -1 (pre-dose), 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of occupancy
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
percentage of occupancy
  Baseline | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0]
  1H | 67.51 [-16.4 to 96.0] | 99.13 [91.9 to 100.0]
  2H | 85.26 [68.5 to 100.0] | 92.53 [88.7 to 100.0]
  4H | 84.93 [76.0 to 100.0] | 92.26 [87.7 to 100.0]
  8H | 87.08 [69.9 to 95.3] | 92.48 [85.0 to 98.7]
  24H | 68.13 [51.5 to 87.9] | 91.32 [82.1 to 97.9]
  48H | 26.50 [-15.6 to 54.1] | 62.34 [52.5 to 79.4]

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ritlecitinib
Description: Cmax is maximum observed plasma concentration. Cmax for ritlecitinib was observed directly from data.
Time Frame: 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: The analysis population included all participants who enrolled and treated with at least 1 concentration measurement of study treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
nanogram/milliliter (ng/mL) | 297.1 (51) | 1275 (20)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Ritlecitinib
Description: Tmax is time for Cmax. Tmax for ritlecitinib was observed directly from data as time of first occurrence.
Time Frame: 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
hour (hr) | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00]

9. Secondary Outcome: Last Quantifiable Plasma Concentration (Clast) of Ritlecitinib
Description: Clast is last quantifiable plasma concentration. Clast for ritlecitinib was observed directly from data.
Time Frame: 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
ng/mL | 4.812 (87) | 4.036 (666)

10. Secondary Outcome: Average Plasma Concentration From Time 0 to 24 Hours (Cav) of Ritlecitinib
Description: Cav is average plasma concentration from time 0 to 24 hours over the 24 hours period. Cav for ritlecitinib was calculated as area under the plasma concentration-time curve from 0 to 24 hours (AUC24) divided by 24.
Time Frame: 0 (pre-dose), 1, 2, 4, 8, 24 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
ng/mL | 28.42 (51) | 144.9 (42)

11. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Ritlecitinib
Description: AUClast is area under the plasma concentration-time profile from time 0 to the time of the Clast. AUClast for ritlecitinib was determined using linear/log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 8, 24, 48 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
nanogram*hour/milliliter (ng*hr/mL) | 651.4 (50) | 3382 (43)

12. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours (AUC24) of Ritlecitinib
Description: AUC24 is area under the plasma concentration-time curve from time 0 to 24 hours. AUC24 for ritlecitinib was determined using linear/log trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 8, 24 hours post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
ng*hr/mL | 681.8 (51) | 3475 (42)

13. Secondary Outcome: Number of Participants With All-Causality and Treatment-Related Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Relatedness to study treatment was assessed by the investigator. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study treatment and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study treatment up to 35 days after the last dose of study treatment (up to 35 days)
Population: The analysis population included all participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
Participants
  Number of Participants with all-causality TEAEs | 3 | 2
  Number of Participants with all-causality SAEs | 0 | 0
  Number of Participants with treatment-related TEAEs | 0 | 0
  Number of Participants with treatment-related SAEs | 0 | 0

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Relatedness to study treatment was assessed by the investigator. Treatment-emergent are events between first dose of study treatment and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs are classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function.
Time Frame: From the first dose of study treatment up to 35 days after the last dose of study treatment (up to 35 days)
Population: The analysis population included all participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
Participants
  Mild (all causalities) | 3 | 2
  Moderate (all causalities) | 0 | 0
  Severe (all causalities) | 0 | 0
  Mild (treatment-related) | 0 | 0
  Moderate (treatment-related) | 0 | 0
  Severe (treatment-related) | 0 | 0

15. Secondary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline Abnormality
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, erythrocyte, platelet, neutrophils, eosinophils, monocytes, basophils, lymphocytes, etc), chemistry (glucose, calcium, sodium, potassium, chloride, total bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, protein, albumin, etc), and urinalysis (glucose, protein, hemoglobin, ketones, nitrite, leukocytes, urine bacteria, etc). Baseline = the pre-dose measurement on Day -1. Laboratory abnormalities meeting pre-defined criteria are reported for this outcome measure. Only those categories in which at least 1 participant had data were reported. ULN=upper limit of normal. LPF=low power field.
Time Frame: From the first dose of study treatment up to 35 days after the last dose of study treatment (up to 35 days)
Population: The analysis population included all participants who took at least 1 dose of study treatment and with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
Participants
  Monocytes/Leukocytes (%) >1.2*ULN | 0 | 2
  Urine Nitrite >=1 | 1 | 1
  Urine Bacteria (/LPF) >20: number analyzed (Participants) | 1 | 1
  Urine Bacteria (/LPF) >20 | 1 | 0

16. Secondary Outcome: Number of Participants With Pre-defined Criteria for Vital Signs
Description: Pre-defined criteria included: 1) Diastolic blood pressure (DBP), a) supine DBP: less than (<) 50 mmHg, b) supine DBP: change of >= 20mmHg increase, c) supine DBP: change of >= 20mmHg decrease; 2) Systolic blood pressure (SBP), a) supine SBP: <90 mmHg, b) supine SBP: change of >=30mmHg increase, c) supine SBP: change of >=30mmHg decrease; 3) Supine pulse rate, a) <40 bpm, b) >120 bpm. mmHg=millimeters of mercury, bpm=beats per minute.
Time Frame: From the first dose of study treatment up to 35 days after the last dose of study treatment (up to 35 days)
Population: The analysis population included all participants who took at least 1 dose of study treatment and who were evaluated against criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
Number analyzed (Participants) | 8 | 8
Participants
  Supine DBP <50 mmHg | 0 | 0
  Supine DBP change >= 20mmHg increase | 0 | 0
  Supine DBP change >= 20mmHg decrease | 0 | 0
  Supine SBP <90 mmHg | 0 | 0
  Supine SBP change >=30mmHg increase | 0 | 0
  Supine SBP change >=30mmHg decrease | 0 | 0
  Supine pulse rate <40 bpm | 0 | 0
  Supine pulse rate >120 bpm | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 35 days after the last dose of study treatment on Day 1 (up to 35 days)
Arm/Group | RITLECITINIB 50 MG CAPSULE | RITLECITINIB 200 MG CAPSULE
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RITLECITINIB 50 MG CAPSULE (N=8) | RITLECITINIB 200 MG CAPSULE (N=8)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT05128058/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT05128058/SAP_001.pdf